CLINICAL TRIAL: NCT06927349
Title: An Non-randomized Open-label, Multicenter Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics, Preliminary Efficacy of BA1301in Participants With Advanced Solid Tumors.
Brief Title: A Trial to Evaluate Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BA1301 in Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Boan Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA1301/CT-CHN-101
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BA1301 (Experimental): BA1301 is administered intravenously once every three weeks.
  Interventions: Drug: BA1301

INTERVENTIONS:
Drug: BA1301 — BA1301 is administered intravenously once every three weeks.

SUMMARY:
This is an open label Phase 1, First in Human trial designed to evaluate the safety, tolerability pharmacokinetics, preliminary efficacy of BA1301 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent and able to follow the trial treatment protocol and visit plan;
2. Age ≥ 18 years old and ≤ 75 years old, male or female;
3. Patients with locally advanced or metastatic malignant solid tumours that cannot be surgically resected as histologically or cytologically confirmed by standard therapy failure or refusal or inability to tolerate standard treatment regimens.
4. Agree to provide archival or fresh tumour tissue for immunohistochemical evaluation for immunohistochemical detection of CLDN18.2 expression.
5. Eastern Cooperative Oncology Group (ECOG) Strength Status Score of 0 or 1.
6. At least one evaluable lesion according to the efficacy evaluation criteria for solid tumours (RECIST1.1).
7. Adequate organ function.
8. Estimated survival ≥ 3 months;
9. Negative blood pregnancy test result for females of childbearing potential at screening.

Exclusion Criteria:

1. Poorly controlled hypertension as judged by the investigator
2. Received any chemotherapy, radiotherapy, targeted therapy, cell therapy, immunotherapy, ADC drug therapy, major surgery, or other anti-cancer therapy within 28 days prior to the first dose of trial drug.
3. Known hypersensitivity to any ingredient of the therapeutic drug used in the study protocol;
4. Positive hepatitis B virus surface antigen (HBsAg) test; Positive hepatitis C virus (HCV) antibody, treponema pallidum antibody, human immunodeficiency virus (HIV) antibody;
5. Pregnant or lactating females, those who have recently planned to become pregnant;
6. Those who have participated in and received any clinical trial drugs (excluding vitamins and minerals) or clinical trial device intervention within 28 days before signing informed consent;
7. Other serious physical or psychiatric illness or laboratory test abnormalities at screening that may increase the risk of participating in the study, or interfere with the results of the study, and patients who, in the opinion of the investigator, are not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) (according to NCI CTCAE 5.0). | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment, up to 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No